CLINICAL TRIAL: NCT04547062
Title: Monocentric Phase 1 Study With Escalation of Doses of Tocilizumab in Combination With Chemotherapy (Idarubicin and Cytarabine) in Patients With Acute Myeloblastic Leukemia (AML) With Poor Prognosis: TOCILAM"
Brief Title: Monocentric Phase 1 Study With Escalation of Doses of Tocilizumab in Combination With Chemotherapy (Idarubicin and Cytarabine) in Patients With Acute Myeloblastic Leukemia (AML)
Acronym: Tocilam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC20_0282; 2020-003209-77 (EudraCT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML il-6 tocilizumab
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Continual Reassessment Method for MTD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tocilizumab — Administration of tocilizumab at day 8 of induction following a classical induction

SUMMARY:
This is a phase 1 dose escalation study testing the addition of an anti-IL6 (tocilizumab) to standard induction chemotherapy for high-risk AML.

DETAILED DESCRIPTION:
Administration of tocilizumab at day 8 of induction following a classical induction using idarubicin 8mg/m2/d for 5 days and cytarabine 100mg/m2/d for 7 days.

ELIGIBILITY:
Inclusion Criteria:

- AML with a poor prognosis defined according to the criteria below: LAM First line: Age <60 years and unfavorable risk according to the 2017 ELN Age> = 60 years old and intermediate or unfavorable risk according to the ELN 2017 LAM in Relapse: whatever the age

* ECOG <= 2
* Patient eligible for intensive chemotherapy
* Informed consent
* Liver function tests: transaminases <3x normal, bilirubin <1.5X normal
* Creatinine clearance> 60ml / min
* LVEF> = 50%

Exclusion Criteria:

* Uncontrolled infection
* Hep B, C, HIV +
* History of diverticulosis / diverticulitis
* No social security or any other scheme
* Pregnant women or patient unable to take contraception(contraceptive pill, abstinence, IUD unauthorized) in case of fertility. A patient who cannot continue contraception for at least 3 months after the last injection of TOCILIZUMAB is not eligible.
* Lactating women
* Minors
* Adults under guardianship, curatorship or legal protection
* Hypersensitivity to one of the active substances or to one of the excipients
* Patients with tuberculosis
* Patients documented with active COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
number of DLT | 45 days

SECONDARY OUTCOMES:
Number of response | 25 months
Percentage of medullary blaste | 24 months
number of days of neutrophil recovery | 30 months
number of days of platelets recovery | 30 months
Number of death | 30 months
number of days between remission and relapse | 30 months
number of days between remission and death | 30 months
number of days between remission and last follow-up date | 30 months
number of days between Day 1 and last follow-up date | 30 months
number of days between Day 1 and death | 30 months
number of days between Day 1 and relapse | 30 months
number of relapse | 30 months
Number of cytokine | 25 months
Number of tocilizumab | 25 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterlin P, Garnier A, Le Bourgeois A, Guillaume T, Le Bris Y, Theisen O, Bene MC, Eveillard M, Rimbert M, Jullien M, Planche L, Gaschet J, Chevallier P. Tocilizumab in combination with a standard induction chemotherapy in acute myeloid leukaemia patients (TOCILAM study): a single-centre, single-arm, phase 1 trial. EClinicalMedicine. 2023 Sep 28;64:102254. doi: 10.1016/j.eclinm.2023.102254. eCollection 2023 Oct. PMID 37786451